CLINICAL TRIAL: NCT05697861
Title: Long-Term Follow-Up of Subjects Treated With NTLA-2001
Brief Title: Long-Term Follow-Up (LTFU) of Subjects Dosed With NTLA-2001
Status: Recruiting | Type: Observational
Sponsor: Intellia Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ITL-2001-CL-999; 2022-003405-30 (EudraCT Number)
Record Dates: First submitted 2023-01-13; First posted 2023-01-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-05

CONDITIONS: Transthyretin-Related (ATTR) Familial Amyloid Polyneuropathy; Transthyretin-Related (ATTR) Familial Amyloid Cardiomyopathy; Wild-Type Transthyretin Cardiac Amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
This is a follow-up study of subjects who received NTLA-2001 in a previous clinical trial as an observational evaluation of the long-term effects of the investigational therapy.

ELIGIBILITY:
Inclusion Criteria:

1. A subject has completed or discontinued from an Intellia-sponsored clinical study in which a complete or partial dose of NTLA-2001 was received.
2. A subject has provided informed consent for the LTFU study.

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participating sites in an Intellia-sponsored clinical study of NTLA-2001.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2038-03 (Estimated); Study Completion 2038-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related SAEs and Protocol-specified AESIs | up to 15 years
  Long-term safety assessment of any treatment-related SAEs and protocol-specified AESIs

SECONDARY OUTCOMES:
PD biomarkers for ATTR including serum TTR and serum prealbumin | up to 15 years
  Long-term assessment of serum TTR and serum prealbumin

CONTACTS AND LOCATIONS:
Locations (4):
- Clinical Trial Site, Paris, France
- Clinical Trial Site, Auckland, New Zealand
- Clinical Trial Site, Umeå, Sweden
- Clinical Trial Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No